CLINICAL TRIAL: NCT03169218
Title: Effects of Mirror Therapy on Pain and Function on Bilateral Carpal Tunnel Syndrom (MTSTC)
Brief Title: Effects of Mirror Therapy on Pain and Function on Bilateral Carpal Tunnel Syndrom
Acronym: MTSTC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Olga Del Pozo Blanco (Other)
Collaborators: Hospital Universitario La Fe (Other); University Rovira i Virgili (Other)
Responsible Party: Sponsor-Investigator, Olga Del Pozo Blanco, Physiotherapist, Hospital de Manises
Organization: Hospital de Manises (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HManises; 2015/0277 (Other: CEIC)
Record Dates: First submitted 2017-05-22; First posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Adult; Chronic pain; Entrapment neuropathy. Carpal tunnel; Exercise therapy; Humans; Neuronal plasticity; Mirror neurons; Pain/cognitive aspects; Physiotherapy; Somatosensory cortex
MeSH Terms: conditions — Carpal Tunnel Syndrome; Chronic Pain; Median Neuropathy | interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mirror therapy group (Experimental): Mirror therapy group: exercises looking at the reflection in the mirror of the hand moving
  Interventions: Other: Mirror therapy
- Placebo group (Placebo Comparator): Placebo group: exercises performed with the mirror turned to avoid the reflection of the hand and looking at the hand that did not remain hidden.
  Interventions: Other: Placebo group

INTERVENTIONS:
Other: Mirror therapy — The treatment proposed for the mirror group consisted of 8 weeks of treatment, performing a series of exercises 2 times a day / 4 times a week. The first 4 weeks the treatment was done in the hospital next to the physiotherapist for 2-3 days a week, and the next 4 weeks the patient performed the exercises following the same guidelines at home.
  Other Names: Mirror visual feedback; Mirror box therapy
  Arms: Mirror therapy group
Other: Placebo group — The treatment was the same than proposed in inference group but with a mirror covered to avoid the reflexion on the hand and looking at the hand that did not remain hidden.
  Arms: Placebo group

SUMMARY:
The purpose of this study was to evaluate pain and function after mirror therapy as well as level of catastrophism in bilateral carpal tunnel syndrome patients

DETAILED DESCRIPTION:
The sample calculation was performed based on the previous pilot study, in which 10 subjects were included. Through this study, a statistically significant effect on the variables analyzed was demonstrated. Therefore, it was determined to duplicate the initial sample to confirm the effect previously studied, assuming losses of 20%. Thus, the value of n for the clinical trial is 20 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Must be signed the informed consent.
* Bilateral carpal tunnel syndrome: clinic and electromiography positive.
* Aged between 18 and 65 years

Exclusion Criteria:

* Patients undergoing surgical intervention of carpal tunnel syndrome in one of two hands
* Unilateral carpal tunnel syndrome
* Patients with chronic pain and / or previous injury (wrist tumor, lymphedema ...) in either hand
* Patients with systemic diseases (diabetes, thyroid ...)
* Patients with pharmacological treatment to take analgesia for any other chronic pathologies
* Subjects who have suffered from a neurological disease that affects the musculoskeletal system
* Mental illness that prevents the compression and / or realization of the study
* Patients with tattoos, scars and / or marks on any of the hands or distal forearm area
* Pregnant women and minors

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
To evaluate changes on pain | Changes in 8 weeks
  Evaluation on pain through McGill Pain Questionnaire This questionnaire is self-administered.

SECONDARY OUTCOMES:
To evaluate changes on the function of the upper limb. | Changes in 8 weeks
  Evaluation on function through disabilities of the arm, shoulder and hand questionnaire (DASH)

OTHER OUTCOMES:
To evaluate catastrophism associated with pain. | Day 0 of the study
  Evaluation through Pain Catastrophizing Scale This questionnaire is self-administered

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Monterde, PT, Phd, Study Director — Faculty of Medicina i Ciències de la Salut; University Rovira i Virgili
Locations (1):
- Hospital de Manises, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lázaro C, Fèlix B, Torrubia R, Baños JE. The development of a Spanish questionnaire for assessing pain: preliminary data concerning reliability and validity. Eur J Psychol assesment. 1994;10(2):145-51.
- [Background] Garcia Campayo J, Rodero B, Alda M, Sobradiel N, Montero J, Moreno S. [Validation of the Spanish version of the Pain Catastrophizing Scale in fibromyalgia]. Med Clin (Barc). 2008 Oct 18;131(13):487-92. doi: 10.1157/13127277. Spanish. PMID 19007576
- [Background] Hervas MT, Navarro Collado MJ, Peiro S, Rodrigo Perez JL, Lopez Mateu P, Martinez Tello I. [Spanish version of the DASH questionnaire. Cross-cultural adaptation, reliability, validity and responsiveness]. Med Clin (Barc). 2006 Sep 30;127(12):441-7. doi: 10.1157/13093053. Spanish. PMID 17040628